CLINICAL TRIAL: NCT01602640
Title: Sedation and Analgesia in Intensive Care: Comparison of Morphine and Fentanyl/Midazolam
Brief Title: Comparison of Morphine and Fentanyl/Midazolam in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Los Andes IPS (Other)
Responsible Party: Principal Investigator, EFRAIN RIVEROS, Principal investigator, Clínica de Los Andes IPS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ANDES001
Record Dates: First submitted 2012-04-18; First posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Respiratory Failure
Keywords: sedation; critical care; morphine; fentanyl; analgesic based sedation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Experimental)
  Interventions: Drug: Morphine infusion
- Fentanyl and Midazolam (Active Comparator): Control
  Interventions: Drug: Fentanyl and Midazolam infusion

INTERVENTIONS:
Drug: Morphine infusion — Conventional dose
  Arms: Morphine
Drug: Fentanyl and Midazolam infusion — Conventional dose
  Arms: Fentanyl and Midazolam

SUMMARY:
Hypothesis: Morphine infusion decreases time to mechanical ventilation weaning and extubation, as compared to the combination of fentanyl and midazolam in critically-ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to ICU requiring mechanical ventilation Informed consent

Exclusion Criteria:

* Less than 18 years old
* Consent denial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time from sedation discontinuation to first T-Tube time from sedation | 12-120 hours

SECONDARY OUTCOMES:
Time from sedation discontinuation to extubation time from sedation | 12-180 hours

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros, Principal investigator, Principal Investigator — Clinica de los Andes IPS
Locations (1):
- Clinica de los Andes IPS, Tunja, Departamento de Boyacá, Colombia